CLINICAL TRIAL: NCT04108234
Title: Safety, Tolerance and Pharmacokinetics of Hydrochloric Acid (R) -Ketamine Nasal Spray in Healthy Subjects: A Randomized, Double Blind, Placebo-Controlled Phase I Clinical Trial
Brief Title: A Study of HR071603(Ketamine Nasal Spray) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR071603-101
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: HR071603 monotherapy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): HR071603,nasal spray,dose escalation.
  Interventions: Drug: HR071603
- Treatment group B (Placebo Comparator): Placebo, nasal spray
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HR071603 — HR071603 monotherapy ,nasal spray
  Other Names: R-ketamine
  Arms: Treatment group A
Drug: placebo — placebo,nasal spray
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the safety and pharmacokinetics of HR071603 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent prior to the start of any activity related to the trial, and have a thorough understanding of the purpose and meaning of the trial and be willing to comply with the protocol;
2. Healthy males aged between 18 and 45 (including both ends);
3. Weight ≥ 50kg, body mass index (BMI) in the range of 18.5 ~ 23.9 (including both ends);
4. During the trial and within 30 days after the administration, willing to take contraceptive measures and ensure that no sperm is donated.

Exclusion Criteria:

1. A subject considered by the investigator to be unsuitable for nasal spray administration;
2. Allergic to any component of the study drug;
3. The underlying disease is not suitable for participation in the trial;
4. 12-lead ECG results in the screening period are abnormal and clinically significant
5. Liver dysfunction;
6. Serum creatinine > 1.2 × ULN during screening period;
7. Screening for infectious diseases screening hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, human immunodeficiency virus (HIV) antibody test positive;
8. Subject has been thoroughly examined, and the results are abnormal and clinically significant;
9. Major operations were performed within 3 months before the screening period.
10. Donate whole blood/plasma within one month before the screening period, or donate whole blood/plasma more than 400 ml within three months before the screening period;
11. Positive urine drug test;
12. The alcohol breath test is positive; or the average daily intake of alcohol exceeds 15g;
13. Nicotine test is positive;
14. History of drug abuse or alcohol abuse;
15. In the past three months, over five cups of coffee or tea per day were consumed in an average;
16. Any prescription drugs, over-the-counter drugs and health products were used within 2 weeks before screening.
17. Participated in clinical trials of any drug or medical device within 3 months before screening ;
18. Any other medical or psychological condition, which in the opinion of the Investigator, might create undue risk to the participant or interfere with the participant's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | Pre-dose to Day8

SECONDARY OUTCOMES:
Assessment of PK parameter-Area under drug-time curve (AUC) | Pre-dose to Day2
Assessment of PK parameter-peak time (Tmax) | Pre-dose to Day2
Assessment of PK parameter-peak concentration (Cmax) | Pre-dose to Day2
Assessment of PK parameter-half-life (t1/2) | Pre-dose to Day2
Assessment of PK parameter-apparent clearance rate (CL/F) | Pre-dose to Day2
Assessment of PK parameter-apparent distribution volume (Vz/F) | Pre-dose to Day2

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing AnDing hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided